CLINICAL TRIAL: NCT01612871
Title: Circulating miRNAs as Biomarkers of Hormone Sensitivity in Breast Cancer? Pilot Study.
Brief Title: Circulating miRNAs as Biomarkers of Hormone Sensitivity in Breast Cancer
Acronym: MIRHO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11SEIN12
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer,; hormonotherapy,; miRNAs,; biomarkers; hormone therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hormone therapy treatment (Experimental): Tamoxifen 20 mg/day, Letrozole 2.5 mg/day, Anastrozole 1 mg/day, Exemestane 25mg/day
  Interventions: Drug: Tamoxifen, Letrozole , Anastrozole, Exemestane

INTERVENTIONS:
Drug: Tamoxifen, Letrozole , Anastrozole, Exemestane — Current first line metastatic hormone therapy treatment in hormone dependent breast cancer :
  Tamoxifen 20 mg/day, Letrozole 2.5 mg/day, Anastrozole 1 mg/day, Exemestane 25mg/day

SUMMARY:
This is a biomedical and prospective study of interventional type. The trial will include 29 patients over a period of 15 months + 24 months of follow up maximum.

The study will be conduct in womens with metastatic invasive breast cancer or locally advanced breast cancer and for which treatment with tamoxifen or anti aromatase (first line hormone therapy for metastatic breast cancer) is indicated.

The main objective of this pilot study is to evaluate the feasibility to detect in the circulating blood of patients, before treatment (T0), the presence of the fifteen tissular microRNAs described in preclinical studies as possibly involved in hormone resistance/sensitivity.

In parallel of the detection of these specific miRNAs, we will conduct a larger scale analysis of circulating miRNAs in these patients before (T = 0) and after one month of treatment (T28).

ELIGIBILITY:
Inclusion Criteria:

1. Women of more than 18 years old (menopausal or not)
2. Women with metastatic invasive breast cancer or locally advanced (without surgical project), for which treatment with tamoxifen or anti aromatase

   +/- LH-RH agonist, is indicated (anti-aromatase prescribed for menopausal womens; tamoxifen prescribed for both menopausal, pre menopausal or not menopausal womens).
3. Cancer hormone-expressing estrogen receptor (ER) and / or progesterone receptor (PR) (>= 10% of tumor cells by IHC technique).

   Cancer HER2 negative.
4. Evaluable disease (measurable according RECIST criteria or not)
5. Any previous adjuvant hormone therapy should be discontinued for at least 21 days.
6. One or two prior metastatic lines of chemotherapy are allowed
7. General status WHO 0-2
8. The women of childbearing age must use an effective contraception for the duration of the study
9. Informed consent obtained and signed before any specific study procedure
10. Patient member in a national insurance scheme

Exclusion Criteria:

1. Patient already treated with hormone therapy or not having stopped the previous adjuvant hormone therapy for at least 21 days.
2. Prescription of chemotherapy and / or other targeted therapy (other than hormone therapy) for the treatment of the breast cancer
3. Any previous hormone therapy for metastatic or locally advanced (without surgical project) breast cancer
4. Known hypercalcaemia before miRNA dosage at T=0 requiring immediate biphosphonate therapy
5. Any other medical or psychiatric condition or severe or chronic laboratory abnormality making the the inclusion of the patient in the study inappropriate in the opinion of the investigator.
6. Patient unable to follow procedures, visits, examinations described in the study.
7. Pregnant women or nursing mothers will not participate in the study.
8. Patients under legal guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-06-27 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2016-01-28 (Actual)

PRIMARY OUTCOMES:
Rates of patients for which specific tissular miRNAs are detected in blood before treatment (D0) | 1 time point (D0) over a period of 39 months
  MiRNAs will be quantified in plasma using qPCR (quantitative Polymerase Chain Reaction) with the kit "miScriptSYBR Green PCR" (Qiagen)

SECONDARY OUTCOMES:
Analysis of the larger-scale circulating miRNAs in plasma of these patients before (D0) and after one month (D28) of treatment with tamoxifen or anti aromatase | 2 time points (D0 and D28) over a period of 39 months (3 years and 3 months)
Correlation between the specific miRNAs initial expression and the appearance of an objective response or clinical benefit of hormone therapy and the time to progression | 39 months (3 years and 3 months)
Rate of objective responses, defined as the number of patients with a complete or partial response. | 39 months (3 years and 3 months)
The time to progression, defined as the time from patient inclusion to the date of the first documented tumor progression | 39 months (3 years and 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Florence DALENCr, PhD, Principal Investigator — Institut Claudius Regaud
Locations (2):
- France (2):
  - Centre Val d'Aurelle - Paul Lamarque, Montpellier
  - Institut Claudius REGAUD Toulouse, Toulouse